CLINICAL TRIAL: NCT03973216
Title: Evaluating a Group-based Therapeutic Yoga Program for Burnout
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 caused the group format to shift, therefore the intervention was not delivered in the same manner as the one described in the proposal. The study was stopped as the intervention may not be delivered as planned even following COVID-19.
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Elizabeth Alvarez, Assistant Professor, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Yoga MD for burnout
Record Dates: First submitted 2019-05-22; First posted 2019-06-04 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Anxiety; Insomnia; Burnout, Professional; Depression; Loneliness
Keywords: Anxiety; Yoga; Mindfulness; Group-based therapy
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Burnout, Professional; Depression

STUDY DESIGN:
Intervention Model Description: This study evaluates the effect of the intervention using a single group, before-after study model. The subjects will be evaluated at baseline and followed longitudinally, until study completion and a long-term followup.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A primary care group-based therapeutic yoga program (Experimental): A primary care care group-based therapeutic yoga program that consists of 9 sessions.
  Interventions: Behavioral: A primary care group-based therapeutic yoga program

INTERVENTIONS:
Behavioral: A primary care group-based therapeutic yoga program — The intervention includes therapeutic yoga training and education sessions on benefits of yoga and effects of stress on the body.

SUMMARY:
This study is evaluating a group-based therapeutic yoga program for burnout. This study aims to understand the feasibility of running the program (i.e. of recruiting participants, the resources required to run the program, etc) and the effectiveness of the program (i.e. in decreasing participants' mental health symptoms).

DETAILED DESCRIPTION:
A primary care group-based therapeutic yoga program, the Yoga MD program, was developed by a primary care / emergency physician practicing in Toronto, Ontario. The program was started in 2014 and is run through a medical centre in Toronto, Ontario. The purposes of the program are to understand:

* key concepts of yoga, mindfulness, compassion, acceptance and how these can help with personal transformation
* how stress is carried in the body (embodiment of stress) and how stress manifests as anxiety, pain, or other symptoms
* what happens when stress accumulates in the body
* the role of self-compassion in the response to stress
* how to cope with difficult emotions that may contribute to stress
* how to deal with difficult people and trying relationships
* the importance of connecting with, and caring for ourselves to reduce accumulated stress
* how to solidify healthier patterns to build resilience to stress faced in daily life.

This study evaluates the 9 weekly sessions using a before-after interventional design. Participants have data collected at baseline, and at 9 weeks and 8 months after the yoga program ends, and changes in mental health outcomes are observed.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18
* Must be enrolled in therapeutic yoga program

Exclusion Criteria:

* no formal exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-30 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder - 7 (GAD-7) | Change from baseline each week until 9 weeks and at 8 months post-baseline
  The GAD-7 is a validated instrument for the diagnosis and treatment response of anxiety disorders (Spitzer et al., 2006; Hinz et al., 2017). It is comprised of 7 questions with 4 answer options, ranging from "not at all" to "nearly every day"and scored 0-3 with a total score ranging from 0-21 (Spitzer et al., 2006). Scores of 5-9, 10-14, and 15-21 represent mild, moderate and severe generalized anxiety disorder, respectively. In the primary care setting, the GAD-7 has high diagnostic validity, with a threshold of 10 exhibiting a sensitivity of 89% and specificity of 82% for generalized anxiety disorder (Spitzer et al., 2006). Other conditions related to generalized anxiety disorder including panic disorder, social anxiety disorder and post-traumatic stress disorder have also been sensitive to a GAD-7 score of 10 (Kroenke et al., 2007).

SECONDARY OUTCOMES:
The Insomnia Severity Index | Change from baseline each week until 9 weeks and at 8 months post-baseline
  The Insomnia Severity Index, a 7-item scale, was identified as the most fitting validated scale to identify insomnia symptoms (Bastien et al., 2001). Each of the questions is measured on a scale of 0-4 and the answers are added up to get a total score.
  Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
The Perceived Stress Scale | Change from baseline each week until 9 weeks and at 8 months post-baseline
  The Perceived Stress Scale contains ten items and is designed to measure the degree to which situations in one's life are appraised as stressful (Cohen, 1994). The minimum score is 0 and the maximum score is 40, with higher scores indicating higher levels of stress.
The Maslach Burnout Inventory | Change from baseline each week until 9 weeks and at 8 months post-baseline
  The Maslach Burnout Inventory is a 22- item scale that is divided into three sub-scales: Emotional Exhaustion, Depersonalization, and Personal Accomplishment. Items are scored using a 7 level frequency scale from "never" to "daily." The 9-item Emotional Exhaustion scale measures feelings of being emotionally overextended. Scores from 0-16 represent low burnout, 17-29 represent moderate burnout, and 30 and over is high burnout. The 5-item Depersonalization scale measures a dehumanization in interpersonal interactions/ Scores of 0-5 represent low burnout, 6-11 represent moderate burnout and 12 or over represent high burnout. The 8-item Personal Accomplishment scale measures feelings of successful achievement in one's work with people. Scores of 33 or less represent high burnout, 34-39 represent moderate burnout, and 40 or over represent low burnout (Maslach, Leiter & Jackson, 1996).
The Adverse Childhood Events (ACE) | Only at baseline
  The Adverse Childhood Events (ACE) Scale includes 10 questions about childhood abuse and exposure to forms of household dysfunction before the age of 18 There is a maximum score of 10, which indicates a greater number of adverse childhood events. The higher your ACE score, the higher your risk of health and social problems (Felitti et al., 1998).
Patient Heath Questionnaire 9 (PHQ-9) for depression | Change from baseline each week until 9 weeks and at 8 months post-baseline
  The Patient Health Questionnaire-9 (PHQ-9) is made up of nine questions and is diagnostic for depression. Importantly, the PHQ-9 has also been found to be sensitive to change for monitoring of treatment outcomes (Kohrt et al, 2016; Lowe et al, 2004). The PHQ-9 asks participants, "Over the last 2 weeks, how often have you been bothered by any of the following problems?" All answers have four options ranging from "not at all," "several days," more than half the days," or "nearly every day" for a number of symptoms related to depression. Major depression and other depressive syndromes are diagnosed based on answers of "more than half the days" or "nearly every day" to "Little interest or pleasure in doing things" or "Feeling down, depressed, or hopeless" plus 2-5 or more of the other symptoms.
The Sheehan Disability Scale | Change from baseline each week until 9 weeks and at 8 months post-baseline
  The Sheehan Disability Scale is a 3-item scale that assesses impairment in three areas: work, social and family (Sheehan, 1983). The questions inquire about the degree to which one's burnout, panic, anxiety, phobia, or depressive symptoms interfere with work/school, social life, and family. The scale ranges from 0 (not at all) to 10 (extremely), with higher scores indicating greater disability. The 3 items can also be summed into a single dimensional measure of global functional impairment that rages from 0 (unimpaired) to 30 (highly impaired).
The short-form Self-Compassion Scale | Change from baseline each week until 9 weeks and at 8 months post-baseline
  The short-form Self-Compassion Scale includes twelve items and is comparable to the longer, 26-item, scale. The short form includes two items each on self-kindness, self-judgement, common humanity, isolation, therapeutic yoga and overidentified items.(Raes, Pommier, Neff, & Van Gucht, 2011). The scale ranges from 1- 5, with 1 indicating almost never, and 5 indicating almost always. Subscale scores are computed by calculating the mean of subscale item responses and total mean scores are also calculated for a total self-compassion score.
The Readiness for Change Scale | Change from baseline each week until 9 weeks and at 8 months post-baseline
  The Readiness for Change Scale contains 3 questions regarding making a change in one's life. It is based on a 10-point scale, and scores range from 0-30. Lower numbers indicate less readiness, and the higher numbers indicate greater readiness for change (Center for Substance Abuse Treatment, 1999).
The DeJong Gierveld 6-item Loneliness Scale | Change from baseline each week until 9 weeks and at 8 months post-baseline
  The DeJong Gierveld 6-item Loneliness Scale captures both emotional loneliness (missing an intimate relationship) and social loneliness (missing a wider social network) (Gierveld et al., 2006; Grygiel et al., 2016). Answer choices include: "Yes", "More or Less", and "No". On the negatively worded items, the neutral and positive answers are scored as "1". Therefore, on questions 1-3 score Yes=1, More or less=1, and No=0. On the positively worded items, the neutral and negative answers are scored as "1". Scores range from 0-6, with higher scores indicating higher levels of loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Alvarez, MD, Principal Investigator — McMaster University; Arielle Sutton, MPH, Principal Investigator — McMaster University
Locations (1):
- Clairhurst Medical Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Hinz A, Klein AM, Brahler E, Glaesmer H, Luck T, Riedel-Heller SG, Wirkner K, Hilbert A. Psychometric evaluation of the Generalized Anxiety Disorder Screener GAD-7, based on a large German general population sample. J Affect Disord. 2017 Mar 1;210:338-344. doi: 10.1016/j.jad.2016.12.012. Epub 2016 Dec 18. PMID 28088111
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Cohen, S. (1994). Perceived Stress Scale. Psychology, 1-3. https://doi.org/10.1037/t02889-000
- [Background] Maslach, C., Jackson, S. E., & Leiter, M. P. (1996). Maslach Burnout Inventory Manual. Evaluating Stress: A Book of Resources. https://doi.org/10.1038/oby.2012.27
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Kohrt BA, Luitel NP, Acharya P, Jordans MJ. Detection of depression in low resource settings: validation of the Patient Health Questionnaire (PHQ-9) and cultural concepts of distress in Nepal. BMC Psychiatry. 2016 Mar 8;16:58. doi: 10.1186/s12888-016-0768-y. PMID 26951403
- [Background] Lowe B, Unutzer J, Callahan CM, Perkins AJ, Kroenke K. Monitoring depression treatment outcomes with the patient health questionnaire-9. Med Care. 2004 Dec;42(12):1194-201. doi: 10.1097/00005650-200412000-00006. PMID 15550799
- [Background] Sheehan, D.V. (1983) The Anxiety Disease. Scribner, New York.
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Gierveld, J. D. J., & Tilburg, T. V. (2006). A 6-Item Scale for Overall, Emotional, and Social Loneliness: Confirmatory Tests on Survey Data. Research on Aging, 28(5), 582-598. https://doi.org/10.1177/0164027506289723
- [Background] Grygiel P, Humenny G, Rebisz S. Using the De Jong Gierveld Loneliness Scale With Early Adolescents: Factor Structure, Reliability, Stability, and External Validity. Assessment. 2019 Mar;26(2):151-165. doi: 10.1177/1073191116682298. Epub 2016 Dec 8. PMID 27932403
- [Derived] Alvarez E, Sutton A, Barton B, Vaidya S. Evaluating a group-based Yoga of Stress Resilience programme: a pragmatic before-after interventional study protocol. BMJ Open. 2020 Mar 31;10(3):e035862. doi: 10.1136/bmjopen-2019-035862. PMID 32234747